Informed Consent Form (ICF) for Study EBS.AVA.212: A Phase 3, Randomized, Double-blind, Parallel-group Trial to Evaluate the Lot Consistency, Immunogenicity, and Safety of AV7909 for Postexposure Prophylaxis of Anthrax in Healthy Adults

ICF Document version / date: Version 2.0 / 29-Jan-2019

NCT number: NCT03877926

# Informed Consent Form to Take Part in a Clinical Research Study and Authorization to Disclose Health information

Sponsor / Study Title: Emergent Product Development Gaithersburg, Inc. / "A

Phase 3, Randomized, Double-blind, Parallel-group Trial to Evaluate the Lot Consistency, Immunogenicity, and Safety of AV7909 for Postexposure Prophylaxis of Anthrax in

Healthy Adults"

Protocol Number: EBS.AVA.212

Principal Investigator:

(Study Doctor)

«PiFullName»

Telephone: «IcfPhoneNumber»

**Additional Contact(s):** 

(Study Staff)

«AdditionalStaffMemberContacts»

Address: «PiLocations»

You are being asked to take part in a research study. This Informed Consent Form will tell you about:

- The study and what will happen to you as a participant in the study,
- Possible benefits and risks to you if you choose to take part in the study, and
- Your rights as a participant in the study.

Before you agree to take part in the study, you must read, sign, and date this Informed Consent Form. Please read this form and ask as many questions as you need to be sure that you understand what will happen to you in this study. You should only sign and date this form if the study doctor or study staff have answered all your questions and you decide that you want to be part of this study. The study doctor or a member of the study staff will also sign and date this form. You will be given a copy of this signed and dated Informed Consent Form to keep. It is your choice to take part in this study because joining this study is voluntary. There will be no penalty or changes to your medical treatment if you choose not to take part in this study. Signature and date on this form does not mean you will automatically get in the study. Only after you sign and date this form can the study doctor do any tests to see if you meet all the requirements to join the study.

Participating in a research study is not the same as getting regular medical care. The purpose of regular medical care is to improve or monitor your health. The purpose of a research study is to gather information about how safe the study drug is and how well it works. Being in this study does not replace your regular medical care.

# **INFORMATION ABOUT THIS RESEARCH STUDY**

#### 1 INTRODUCTION

This study is being paid for by the Biomedical Advanced Research and Development Authority (BARDA; part of the United States [U.S.] Department of Health & Human Services) together with a company called Emergent Product Development Gaithersburg, Inc, hereafter called "Emergent." Emergent is the sponsor of this study and makes the study drug being tested, a study vaccine called AV7909. AV7909 study vaccine is being studied to see if it can prevent anthrax disease.

#### 1.1 What are Vaccines?

Vaccines are given to people to prevent them from getting a specific infection or disease by helping their immune system to fight off the bacteria or virus that causes the infection or disease. The immune system is the body's natural defense against germs and other invaders. Through a series of steps called the immune response, the immune system attacks germs that invade your body and cause disease. Vaccines help the immune system make special proteins called antibodies that can help fight an infection at a later point in time. This may result in a milder infection (you get better sooner) or even keep you from getting sick at all after being exposed to the bacteria or virus at a later point in time.

#### 1.2 What is Anthrax Disease?

Anthrax is a disease that can affect both animals and humans. It is caused by the bacteria called *Bacillus anthracis* (also written as *B. anthracis*). Though very rare, people can get anthrax from direct skin contact from infected animals, wool, meat, or hides; breathing or ingesting the bacteria, or by injection (through a shot). Anthrax is usually a skin disease that causes open sores on the skin and usually fever and tiredness. Two out of ten people who catch the skin type of anthrax die if they do not receive treatment. When *B. anthracis* is breathed in, the resulting disease is much more serious than the skin disease. The first symptoms may include a sore throat, mild fever and muscle aches. Within several days, these symptoms are followed by severe breathing problems, shock, and often meningitis (inflammation of the membrane that covers the brain and spinal cord). Once symptoms appear, most people who catch this form of anthrax die even if they are treated with antibiotics.

# 1.3 What is AV7909 Study Vaccine?

AV7909 study vaccine is made up of the same drug substance found in an approved vaccine called BioThrax\*. BioThrax vaccine, which is also made by Emergent, is a Food and Drug Administration (FDA) approved vaccine used to prevent anthrax infection in adults who are at high risk of getting anthrax (such as certain people in the military). BioThrax vaccine helps people make antibodies against the bacteria that cause anthrax. AV7909 study vaccine also contains another substance called CPG 7909 (not found in BioThrax) that works by boosting the vaccine's effects to increase the body's immune response. Being a combination of BioThrax plus CPG 7909, it is believed that AV7909 study vaccine can work just as well if not better than BioThrax vaccine to help the body make antibodies against the bacteria that cause anthrax.

The use of AV7909 study vaccine is "investigational," meaning the study vaccine has not been approved for sale in the U.S. by the FDA. The study doctor is being paid to conduct this study.

# 1.4 What is the Purpose of this Study?

The purpose of this study is to see if the AV7909 study vaccine is safe, if it produces any side effects, and to measure the body's immune response to AV7909 study vaccine. This study will also test if three different lots of the AV7909 study vaccine (meaning three different batches of the study vaccine made at different times using the same manufacturing process) result in generally the same amount of antibodies being made by the body.

Researchers want to find out if AV7909 study vaccine can help protect against the bacteria that causes anthrax. They will test if the AV7909 study vaccine works by looking for antibodies (natural immune proteins) in your blood several times after you receive the study vaccine. You will NOT come into contact with the anthrax bacteria as part of this research study; therefore, you will NOT be at risk of anthrax infection.

# 1.5 What is this Study About?

Approximately 3,850 healthy participants who are between 18 and 65 years old will be enrolled in this study in about 40 medical clinics across the U.S. Some people will receive AV7909 study vaccine (investigational vaccine) and some will receive BioThrax vaccine (FDA-approved vaccine). This study is "double-blind," which means that you and the study doctor will not know which study vaccine you are receiving (AV7909 study vaccine or BioThrax vaccine). This is done so that you and the study doctor won't accidentally influence the study results either in a good way or a bad way by knowing ahead of time what study vaccine you've been given. AV7909 study vaccine is given as two shots separated by two weeks while BioThrax vaccine is given as three shots each separated by two weeks. To ensure you and the study doctor don't guess which vaccine you are getting because of a difference in the number of shots given, the people getting AV7909 study vaccine will receive two shots of AV7909 study vaccine followed by a third shot of placebo, which is a dummy shot consisting of sterile salt water with no medication in it. This third shot of placebo will be given two weeks after the second dose of AV7909 study vaccine.

Be aware that this form refers to AV7909 vaccine, BioThrax, and placebo as "study shot" because a vaccine is given as a shot in the arm.

#### 2 ELIGIBILITY

# 2.1 Who can participate in the study?

People who served in the U.S. military after 1990 cannot participate in this study because they may have already received the BioThrax vaccine. In addition, if you plan to enlist in the military within 15 months after joining the study, you cannot participate in the study. If you are considering enlisting in the military, please tell the study doctor.

In order to be in this study, you must additionally meet the following requirements:

- Sign and date this Informed Consent Form
- Be 18-65 years old and in good health, with no recent signs (within the past five years) of drug or alcohol abuse
- Have a Body Mass Index (BMI) less than or equal to 35.0 kg/m<sup>2</sup> (the study doctor will measure your height and weight to determine your BMI)
- Be able to have blood drawn without too much difficulty
- For women able to have children:
  - Have negative pregnancy tests before enrolling in the study and before getting your first study shot
  - Not be currently breast-feeding
  - Have no intention to become pregnant at any time while participating in the study
  - Use an acceptable form of birth control to prevent pregnancy at least 1 month prior to Study Day 1 through Month 13

An acceptable form of birth control for women is any of the following:

- 1) No sexual intercourse;
- 2) Previous bilateral tubal ligation procedure (tubes tied);
- 3) Monogamous relationship with a vasectomized partner (vasectomy performed at least six months ago); or
- 4) Any of these forms of birth control: pill, intrauterine device (IUD), implantable or injectable contraceptive (for example, Norplant® or Depo-Provera®), removable device (for example., NuvaRing® or Evra® patch), or double-barrier method (condom with spermicide, diaphragm with spermicide).

The study doctor or study staff will ask you about your preferred birth control method and review it with you at every study visit or phone call.

- Have no plans to receive a vaccine shot (for example, flu vaccine, tetanus vaccine) from seven days before your first scheduled study shot through 2 weeks after receiving your final study shot
- Take no medications before or during the study that your study doctor determines could affect your body's immune response
- Have not previously had anthrax disease, or been exposed to anthrax, or previously received a shot of anthrax vaccine
- Have not previously had a severe allergic reaction to a vaccine, and have no known allergy to synthetic oligonucleotides, aluminum, formaldehyde, benzethonium chloride (also called phemerol), or latex
- Have no plan for elective surgery at any time while participating in study

- Have no tattoo/scar/birthmark or any other skin condition affecting the upper arm areas where the study shot will be given
- Not be participating in any other research study in which you receive an investigational product (meaning it is not FDA-approved) at the same time as this study

Tell the study doctor if you don't meet one or more of these study requirements. Before you can be enrolled in the study, the study doctor will perform a physical examination, run some laboratory tests, and ask you some questions about your health and medical history (refer to Section 4 of this Informed Consent Form). Based on the results, the study doctor will decide if you qualify for participation in the study.

#### 3 PARTICIPANT RESPONSIBILITIES

# 3.1 What will happen while on the study?

You will be expected to attend all planned visits and accept all study-related phone calls as listed in the study treatment schedule described in Section 4 of this Informed Consent Form. You must additionally:

- Show up on time for all five scheduled study visits. Alert the study doctor/study staff as soon as possible if you must reschedule a visit for any reason.
- Allow the study doctor/study staff to draw blood and take urine samples on the study days listed in this Informed Consent Form.
- Tell the study doctor/study staff about all past and current medical conditions for which you have received medical care or treatment.
- Tell the study doctor/study staff about any past (within 30 days before your first study visit) or new medications you are taking.
- Tell the study doctor/study staff if you do not feel well or notice unusual changes in your mind or body while in the study.
- Allow the study staff to give you a study shot in the arm on Study Day 1, Study Day 15, and Study Day 29.
- When at home, complete an electronic diary (e-diary) once a day for at least one week after
  each study shot to describe your study shot-related symptoms. If you don't have a personal
  smartphone, tablet, or computer with internet access to do this, the study staff will loan you a
  mobile device, to be used only for purposes of this study and to be returned to study staff when
  directed.
- If you are a woman able to have children, use an acceptable method of birth control (refer to Section 2) for the duration of the study and let the study doctor/study staff know immediately if you know or think you may be pregnant or when there has been a change in your method of birth control.
- Agree not to receive any commercially available shot such as a flu shot, until at least 2 weeks after the last study shot.

- Agree not to take certain medications used to treat fever or muscle aches during the 24 hours before and 24 hours after receiving the study shot, because these medications may hide the side effects of the study shot. This includes any aspirin- or Tylenol-containing medications and any non-steroidal anti-inflammatory medications such as ibuprofen, naproxen, diclofenac and celecoxib.
- Respond to the study doctor/study staff when they call you about 3, 6, 9, and 12 months after
  the last planned study shot to find out about any changes to your general health since the last
  study visit or phone call.
- Agree to come to the study doctor's office when requested by the study doctor or study staff
  outside of a scheduled study visit or phone call in order to undergo a medical evaluation and
  blood/urine tests if necessary.

#### 4 STUDY TREATMENT SCHEDULE

If the study doctor says you can be in the study and you agree to participate, your time in the study will last about 15 months. You will have to come to the study doctor's office about five times during the first 3 months of the study. The study staff will tell you when to come in for your study visits. On each of the three visits that you receive the study shot, the visits may last about 2 to 3 hours each. The rest of your study visits may last about 1 to 2 hours each. At the end of all the study visits, you will receive phone calls from the study doctor/study staff spaced several months apart over 12 months so they can check up on your health and well-being. See below for more information about which tests and procedures will be done at each study visit or phone call and be sure to ask the study doctor or study staff if you have any questions.

# 4.1 Visit 1: Screening Visit (Day -28)

If you agree to participate in the study, you will sign and date this Informed Consent Form before any study procedures are done.

First, a screening visit will be conducted. During this first study visit, the study doctor and/or study staff will collect some information about you and do some tests to find out if you can be in the study. They will:

- Assign you a subject code number that will identify you for the study purposes so that information collected about you is kept private (also see Section 7).
- Ask questions about you (age, sex, race and ethnicity) and your medical history, including
  medicines you take and shots you have had. You will need to tell study staff if you take any
  over-the-counter or prescription medicines and any vitamins or herbs.
- Review the conditions for being in the study with you.
- Perform a complete physical exam.
- Measure your height, weight, and vital signs (blood pressure, temperature, heart and breathing rates).
- Draw blood for some tests (about 3 teaspoons of blood will be collected). You will be tested for signs of illness or infection, including for HIV (human immunodeficiency virus), hepatitis B and

hepatitis C. If you test positive for HIV, hepatitis B, hepatitis C or certain other illnesses or infections, you cannot be in the study. Depending on state law, you may have to sign and date a separate Informed Consent Form before this testing can start. The study doctor or study staff will tell you if the test results are positive. If required by state law, the study doctor or study staff may report a positive test result to the local health department.

- Collect a urine sample to test for signs of illness or infection and for illegal drugs. If your urine
  test shows illness, infection or illegal drugs, you will be told the results and you will not qualify
  to be in the study.
- If you are a woman who is not surgically sterile, draw blood for a pregnancy test (less than a teaspoon of blood will be collected). The study doctor or study staff will tell you if the pregnancy test results are positive; results of the pregnancy testing must be negative in order for you to be in the study. Pregnant women and women who are not using an acceptable form of birth control cannot be in the study. If you have not had a period for more than 12 months in a row, blood will be drawn and tested to verify if you are postmenopausal. Once you are confirmed to be postmenopausal, you will not need to have any more pregnancy tests for the rest of the study.

If you meet the conditions to be in the study, your first study shot will be given within 28 days after this screening visit. The study doctor/study staff will tell you when to come back for your second visit.

# 4.2 Clinic Visits 2 (Day 1), 3 (Day 15), and 4 (Day 29): Study Shot Visits

At your second visit, the study doctor will review with you the conditions for being in the study. If you meet all requirements, the study doctor will enroll you in the study by assigning you by chance (like flipping a coin) to one of the four study groups. You will be in one of the following study groups:

- AV7909 study vaccine Batch 1
- AV7909 study vaccine Batch 2
- AV7909 study vaccine Batch 3
- BioThrax vaccine

Your chances of being assigned to one of the three AV7909 groups versus the BioThrax group will be 6 to 1. Regardless of which group you are in, you will receive 3 study shots in the upper arm during the study, each shot given two weeks apart. The first study shot will be given during your second visit (also called Study Day 1). The second study shot will be given during your third visit, about 2 weeks after the first study shot (called Study Day 15). Your third study shot will be given during your fourth visit, about 4 weeks after the first study shot (called Study Day 29). At the third and fourth visits, you will get the shot in the opposite arm from the one used the last time you got a shot.

At the three study visits when you get study shots (Study Days 1, 15, and 29), the study doctor or study staff will perform the following before you get the study shot:

Review the conditions for being able to receive a study shot on that day (for example, you can't
have a fever or be pregnant).

- Collect urine for a pregnancy test and confirm your method of birth control, if you are a woman who could become pregnant. If this test is positive, blood will be drawn for a more accurate pregnancy test. You will be told the results of this test.
- Review and update your medical history (happens on Study Day 1 only).
- Review how you have been feeling since your last visit.
- Perform a physical exam related to your symptoms, if you have any, and measure your vital signs (blood pressure, temperature, heart and breathing rates).
- Draw blood (about 1½ teaspoons of blood will be collected) to check for substances made by your immune system called antibodies happens on Study Day 1 and Day 29 only).
- Draw blood (about 2 teaspoon of blood will be collected) and collect urine for laboratory testing (happens on Day 29 only). Your blood and urine will be tested for signs of illness or infection.
- Review any medicines you have taken since the last visit.

If you still qualify for receiving the study shot after all of these tests and examinations, you will be given a study shot. Both you and the study doctor will not know what shot you have been given, because another study staff member at the study doctor's office (not the study doctor) will prepare and give you your study shot.

#### After the study shot:

- The study doctor and study staff will check up on you in the study clinic for at least 30 minutes after the study shot to see if you have any reaction to it and also measure your vital signs about 30 minutes after the study shot.
- On Study Day 1, you will be given instructions on how to complete an e-diary on the internet. The e-diary is used to record some types of side effects related to the study shot you may have over the next seven days and any medications you are taking. You will complete an e-diary once a day for seven days after each study shot. If you still have side effects related to the study shot after seven days, you will continue to complete the e-diary until you've had no more symptoms for at least two days in a row. To help you complete the e-diary, you will be given a thermometer to record your temperature. You will also be given a measuring tool and shown how to measure the size of any redness or swelling on your arm where you received your study shot. If you need a mobile device in order to access the e-diary, one will be loaned to you by the study staff to be used for the purposes of this study.
- If you previously completed an e-diary, the study doctor or study staff will review it with you.
- Any side effects will be recorded by the study doctor.
- The next study visit will be scheduled.

#### 4.3 Last Clinic Visit

At the fifth and final study visit (Study Day 64), the study doctor or study staff will do some or all of the following:

- Review how you have been feeling since the previous visit. Any side effects will be recorded by the study doctor.
- Perform a complete physical exam and measure your vital signs (blood pressure, temperature, heart and breathing rates).
- Draw blood to check for substances made by your immune system called antibodies (about 1½ teaspoons of blood will be collected).
- Draw blood (about 2 teaspoons of blood will be collected) for laboratory testing. Your blood will be tested for signs of illness or infection.
- In women who are able to have children, draw blood) less than a teaspoon for a pregnancy test and confirm your method of birth control. You will be told the results of this test.
- Review any medicines you have taken since the last visit.
- Collect the mobile device provided to you for e-diary entry (if not already returned to the study staff).

# 4.4 Early Withdrawal Visit

You can withdraw from the study at any time without penalty. The study doctor may also decide you can't receive any more study shots (for example, if you have an allergic reaction to the study shot, or you have a fever on a day when you were supposed to receive a study shot, or you become pregnant). Once you've received at least one study shot and either you or the study doctor decides you can't receive any more study shots, you will continue with your scheduled study visits and study follow-up phone calls. You will have the tests and procedures described in Section 4. However, you won't have any more study shots and may not have any more blood samples collected to test the amount of antibodies that could protect you against anthrax. This will allow the study doctor and study staff to check up on your health and well-being for the entire study length.

If, however, you choose not to be in the study anymore and have not yet reached your fifth study visit (Study Day 64), the study doctor/study staff will ask you to come to the doctor's office for a final visit (called an Early Withdrawal Visit) to check your health one last time.

At the Early Withdrawal Visit, the study doctor or study staff will do some or all of the following:

- Review how you have been feeling since the previous visit. Any side effects will be recorded by the study doctor.
- Perform a complete physical exam and measure your vital signs (blood pressure, temperature, heart and breathing rates).
- Review any medicines you have taken since the last visit.
- In women who are able to have children, draw blood (less than a teaspoon) for a pregnancy test and confirm your method of birth control. You will be told the results of this test.
- Draw blood (about 2½ teaspoons of blood will be collected) and collect urine for laboratory testing. Your blood and urine will be tested for signs of illness or infection.

- If you withdraw before study Day 29, you may be asked to draw blood to check for substances made by your immune system called antibodies (about 1½ teaspoons of blood will be collected).
- If you recently completed an e-diary, review it with you.
- Collect the mobile device provided to you for e-diary entry (if not already returned to the study staff).

# 4.5 Phone Calls at Day 43, Months 4, 7, 10, and 13

You will receive phone calls from the study doctor or study staff at Day 43, Months 4, 7, 10, and 13, which will occur, respectively, about 2 weeks, 3 months, 6 months, 9 months, and 12 months after you receive your last scheduled study shot. You will be asked about your e-diary entries (at Day 43 only). You will also be asked about your health since your last visit or the last time you received a phone call. If you are a woman who could have children, you will be asked to confirm your method of birth control. You may also be asked about any medications you have taken. The study doctor may ask you more detailed questions about any side effects and possibly refer you to a specialist if more tests are needed. The study doctor may ask you to come to the study doctor's office to collect blood in order to test it for antibodies that may indicate an autoimmune response.

# 4.6 What will happen to any samples you give?

## Samples collected for safety:

Blood and urine samples will be collected from you for safety testing. These samples will be kept until testing is completed or until the sample is no longer usable. The samples will then be destroyed. These samples will be labeled with your subject code number and will not contain your name or any other personal information.

#### Samples collected for future use:

If you agree, samples of your blood will be stored for possible future re-testing as part of continued research on the anthrax vaccine. Any blood samples left over from the immune response testing will be stored frozen at a long-term storage facility. You will not be asked to provide additional blood samples.

Samples may be stored until at least 2 years after the last marketing application is approved (AV7909 is not approved for sale), or is no longer pending, or the investigation of AV7909 is discontinued.

These samples will only be used for research purposes and will not be sold or used directly for the production of commercial products.

Allowing retention of your leftover blood samples for future research is optional. You will be asked to agree or decline to the retention of your leftover blood samples at the end of this form.

Identifiers will be removed from your private information (personal and health information collected as part of this study) and any biospecimens (blood samples). These samples will be labeled with your subject code number and will not contain your name or any other personal information. After the information or biospecimens can no longer be readily identified as yours, it may be used for future research studies or sent to another investigator for future research studies. You will not be asked to provide additional informed consent for such use.

Medical research from your blood samples may result in new products or discoveries. These may have value to others but you will not share in any financial or other benefits from the use of your blood samples.

You will not be informed if clinically relevant information (information that can be used to support the health care of people) is discovered during research using your samples.

#### 5 RISKS AND BENEFITS

# 5.1 What are the Risks of Being in this Study?

All medicines may cause side effects. There may be side effects of AV7909 or BioThrax vaccines that are not yet known. AV7909 has been previously studied in people. AV7909 has already been given to about 241 people in 3 completed studies.

The known side effects are listed below. By agreeing to take part in this study, you should know that you might experience any of the problems listed below or other side effects that are not known yet.

# 5.2 What are the possible side effects with AV7909 or BioThrax Vaccines?

The potential side effects listed below, whether related or not to AV7909 were reported during 3 completed clinical studies. These potential side effects may include but are not limited to:

- Reactions on your upper arm where you got the study shot, such as swelling, tenderness, redness, warmth, itching, bruising, bleeding darker skin color, a hardened bump or lump, rash, limited arm movement, pain, burning sensation, or numbness/tingling
- · Feeling very tired all over
- Headache, migraine
- Flu-like symptoms such as fever, chills, and muscle aches
- Decreases or increase in cell blood numbers, such as in the number of white blood cells
- Cold with stuffy nose
- Rapid or fast breathing
- Nausea
- Diarrhea
- Excess gassiness or flatulence
- Toothache
- Vomiting
- Flushing
- Night sweats
- Cough
- Nasal congestion or sore throat

- Upper respiratory tract infection
- Urinary tract infection
- Vaginal infection
- Increased level in liver function tests
- Changes in blood pressure
- Decreased appetite
- Increased glucose
- High or low blood sugar levels
- High or low potassium levels
- High or Low magnesium blood levels
- Difficulty sleeping
- Blood protein or white blood cells in the urine
- Inflammation of voice box
- Slow or fast heart beat (pulse)
- Decreased hemoglobin (eg, anemia)
- Increased level of bilirubin in the blood
- Decreased kidney function
- Abnormal size or change in shape or feel of lymph nodes
- Feeling of body temperature change
- Feeling unwell
- Stomach flu
- Hives
- Numbness and tingling
- Pain [eg, in muscles, joints, jaw, back, neck, chest (non-cardiac), abdomen, ear]
- Skin mole
- Muscle cramps
- · Discomfort in the armpit area
- Indigestion

Sometimes people may have allergic reactions to AV7909 or BioThrax vaccines. If you have a very bad allergic reaction, you could die. Some things you may have during an allergic reaction are:

- A rash
- Having a hard time breathing

- Wheezing
- Sudden drop in blood pressure (making you feel dizzy or lightheaded)
- Swelling around the mouth, throat, or eyes
- Fast pulse
- Sweating
- Nausea
- Hard or fast heart beat or skipping heart beat(s)

Possible risks associated with getting any shot are:

- Dizziness/fainting
- Pain associated with the needle stick
- Nerve or blood vessel damage
- Infection
- Sterile abscess, which is a sore at the point of injection, can be painful and warm to the touch

You should get medical help and contact the study doctor or study staff if you have any of these or any other side effects during the study. Contact information for the study staff can be found on page one of this Informed Consent Form.

AV7909 and BioThrax vaccines are not recommended for anyone who previously had a severe allergic reaction to a vaccine. If you have had a bad allergic reaction to a vaccine in the past, please tell the study doctor. If you are allergic to latex, you cannot participate in this study because the lid on the vaccine container contains a dry natural rubber that could cause an allergic reaction. If you are allergic to latex, please tell the study doctor.

One of the possible risks from one of the substances in the AV7909 study vaccine is overstimulation of your body's immune response, which could result in a chronic autoimmune disease. Chronic means a disease that continues for a long time. An autoimmune disease develops when your immune system, which defends your body against disease, decides your healthy cells are foreign. As a result, your immune system attacks healthy cells. Depending on the type, an autoimmune disease can affect one or many different parts of your body. Because of this possible risk, the study doctor and study staff will check up on your medical condition throughout this study up through 12 months after the last scheduled study shot.

During this study you will be observed for any bad or harmful effects. The study doctor will decide if it is safe for you to keep taking part in the study. Tell the study doctor or study staff right away if you have any problems with your health or the way you feel during the study, whether or not you think these problems are related to the study shots.

It is possible that you could have side effects to AV7909 study vaccine that nobody knows about yet, which could even include death. If the study doctor learns any new information about AV7909 that might change your mind about continuing in the study, the study doctor or study staff will tell you about it in a timely manner.

«PiFullName»

It is possible that receiving AV7909 with your regular medications or supplements may change how AV7909, your regular medications, or your regular supplements work. It is very important that you tell the study doctor about all medications or supplements you are taking during the study and any changes in your overall health.

# 5.3 What are the Possible Risks to Reproduction or to the Unborn Baby (Fetus or Embryo) or Nursing Infant?

If you are pregnant or nursing a child while receiving AV7909 study vaccine, there may be risks to your unborn baby or nursing child. It is not known what these risks are right now.

AV7909 study vaccine and BioThrax vaccine have not been tested in pregnant women or women who are breast-feeding. As a result, pregnant or breast-feeding women are not allowed to join the study. Also, women who want to become pregnant at any time while on the study will not be allowed to join the study. Women who join the study but are able to have children must use an acceptable form of birth control to prevent pregnancy at least 1 month prior to Study Day 1 through Month 13 (after the last study phone visit). See Section 2 of this Informed Consent Form for what is considered an acceptable form of birth control. Be aware that you can still become pregnant even if you use an acceptable birth control method.

If you join the study and are a woman who could get pregnant: The study doctor will ask about your method of contraception and also give you a pregnancy test before you join the study and during every study visit. If you become pregnant during the study or think you may be pregnant, you must immediately tell the study doctor/study staff so that the pregnancy can be confirmed with a blood test and the study doctor knows to stop giving you any more study shots. The study doctor will check up on your health and well-being for the length of the study, and, after the birth, also confirm the health and well-being of your child. If you choose to leave the study early, or even if you complete the study as scheduled but have not yet given birth, the study doctor/staff will contact you at the time of your labor/delivery to check up on your health and also 28 days later to check up on the health of your child.

# 5.4 Are there any other risks?

#### Are there any risks from blood collection?

Some people have discomfort or pain when blood is collected. Some people feel faint or pass out during or shortly after blood is drawn. If you feel faint, lie down right away so you don't get hurt from a fall and tell the study personnel right away. There is a risk of infection, bleeding, swelling, and/or bruising at the spot where blood was taken or a clot may form when blood is collected.

Over four or more study visits, you will give a total of about 13 teaspoons of blood, or less than 1 cup (65.5 mL). For comparison, this is less than half the standard blood donation of about 2 cups (473 mL).

#### Are there any risks of injury that could result from participating in the study?

All forms of medical health diagnosis and treatment – whether routine or experimental – involve some risk of injury. There may also be risks in this study that we do not know about. Even with all the care that is taken, you may still develop medical complications from being in this study. If during this study you get hurt or sick or have any side effect to the study vaccine or study procedure, please contact the

study doctor. If such complications happen, the study doctor will help you get the proper medical treatment.

In the event of an injury that occurs to you as a result of receiving AV7909 study vaccine or BioThrax vaccine or undergoing study procedures, you will receive the necessary medical treatment. In the event that you suffer injury as a direct result of participating in this study, Emergent will cover the costs of reasonable necessary medical treatment not covered by your medical or hospital insurance or by third-party or governmental programs providing such coverage. Emergent or the study doctor will not cover costs for medical care for injuries or illnesses that are not a direct result of study activities. There are no plans to provide other compensation from Emergent or the study doctor.

You are not prevented from seeking to collect compensation for injury related to malpractice, fault, or blame on the part of those involved in the study, including the study clinic or Emergent.

By signing and dating this Informed Consent Form, you do not give up your legal right to look for and receive required medical treatment. You do not give up any rights to seek payment for personal injury by signing and dating this form.

# Are there any benefits to being in the study?

This study is for research purposes only. There is no direct benefit to you from your participation in the study. Information from this study might help researchers develop a new vaccine to prevent anthrax, new tests, or other medications that could help others in the future.

# 6 ALTERNATIVE COURSES OF TREATMENT AVAILABLE (OR ALTERNATIVES TO BEING IN THE STUDY)

The study shot in this study is not being given to you to treat or prevent anthrax or any disease. The other option available to you is not to be in this study.

#### 7 USE OF STUDY RESULTS AND CONFIDENTIALITY OF MEDICAL RECORDS

Your medical and treatment history will be recorded for study purposes. Any information learned about you in this study will be kept private. The study doctor, study sponsor (Emergent), third parties working on behalf of the study sponsor (including BARDA), the ethics board (IRB), and the proper national and international regulatory authorities such as FDA will be able to see your health records and test results to confirm the study data and the safety of study participants. They may copy information from your health records. Your records will be protected and kept as private as possible under local/national/international regulations. By signing and dating this Informed Consent Form, you are granting direct access to these records and test results. Subject to applicable laws, any report that is written about this study will not reveal your identity. If the results of this study are given to medical journals, your identity will not be revealed.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### 8 AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION

Privacy rights of people participating in clinical research studies are protected under the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Your rights as a subject under this act include deciding who has access to your personal health information (called "Protected Health Information").

Protected Health Information is medical information about you that includes your entire historical medical records, all study doctor visits, evaluations, biospecimens (for example, blood samples), laboratory tests, diagnostic tests, procedures, treatments, medications taken, hospitalizations, etc. The study doctor may also get information about your past, present and/or future physical or mental health and/or condition from your primary care doctor. Protected Health Information contains identifiers that can link your medical records specifically to you, such as:

- Your name,
- Your address,
- Date of birth,
- Social security/insurance number,
- Dates and results of various tests and procedures,
- Basic demographic information (such as age, gender, ethnicity/race).

The study information sent to the sponsor and their representative(s) by your study doctor and/or study clinic will not include your name, address or social security/insurance number. As a safety measure to help keep confidentiality, your initials and a subject code number will be used to identify you.

The study doctor will keep this personal health information in your study-related medical records (that we will refer to as "your records") during the study and for 2 years after the last marketing application is approved, is no longer pending, or investigation of AV7909 is discontinued.

By signing and dating this authorization form, you are allowing the study doctor and/or study clinic to have direct access to your Protected Health Information collected in this study, and to receive your Protected Health Information from either your physician or the facilities where you have received health care.

Information collected about you during this study will be used to confirm the safety and effectiveness of AV7909 study vaccine, and the study information may be published in a scientific article. You will not be personally identified in these instances. In addition, the sponsor may re-analyze the results at a later date and combine them with results of other studies.

Your signature and date on this Informed Consent Form authorizes:

 The researchers, study doctors, and/or institution to have access to your Protected Health Information collected as part of this study;

«PiFullName»

- The study doctor and/or institution to receive your Protected Health Information from your physician and/or facilities where you have received any health care;
- Your Protected Health Information to be shared with other persons or organizations involved in the conduct or oversight of this research study, including but not limited to: U.S. Food and Drug Administration (FDA); Biomedical Advanced Research and Development Authority (BARDA); Centers for Disease Control & Prevention (CDC); the IRB used by your study doctor's office; regulatory agencies in other countries; the sponsor and third parties working on behalf of the sponsor; and the laboratory(ies) handling the lab specimens for this study. The other persons and/or organizations need to see your personal health information so they can review the data and to confirm the quality of the study conduct and/or the data collected. These other persons and/or organizations may or may not have the same obligations as the study doctor or institution to protect your Protected Health Information.

The IRB used by your study doctor's office may review your Protected Health Information.

Your Protected Health Information will not be used or given to any other person or entity, except as required by law, or for authorized oversight of this research study. Your Protected Health Information will be used for as long as the sponsor reports study information to the FDA or other countries' regulatory agencies.

You may cancel this authorization in writing at any time by contacting the study doctor listed on the first page of this Informed Consent Form. If you cancel the authorization, continued use is permitted for the Protected Health Information obtained before the cancellation, if its use is necessary in completing the research, including samples collected for future research, if you have agreed to the storage of your leftover blood samples.

If you refuse to provide this authorization, you will not be able to participate in the research study. If you cancel the authorization, then you will be withdrawn from the study.

Finally, federal regulations allow you to obtain access to your Protected Health Information collected or used in this study. However, in order to complete the research study, your access to this Protected Health Information may be temporarily suspended while the research study is in progress. When the study is completed, your right of access to this information will be reinstated.

This authorization will expire once there is no longer a need to review and analyze the information related to this study. Your authorization for the use of your Protected Health Information will not expire, but once the study is over there will be no access or link to your Protected Health Information for anything other than this study. In California and any other state that requires an expiration date, the Authorization will expire 50 years after you sign this authorization document.

| | / | : |
|--------------------------------|-------------|-------------------|
| Signature of Participant | YYYY/MMM/DD | Time (24hr clock) |
| Print Name of Participant Here | | |

#### 9 COSTS AND SUBJECT COMPENSATION

Study shots will be provided by the sponsor. There is no cost to you for any of the study visits or tests.

While you are in the study, you still need to get regular medical care as you normally would seek that care. You (and/or your health care payer) will still have to pay for the costs of your regular medical care that are not a part of this study.

You will receive up to \$\_\_\_\_\_ for each completed study visit and \$\_\_\_\_\_ for each follow-up phone call for a total of \$\_\_\_\_\_. This includes reimbursement for your time and also covers any reasonable travel expenses directly related to the study visits. You will be paid after each visit.

# 10 RIGHT TO ASK QUESTIONS AND/OR WITHDRAW FROM THE STUDY

Your participation in this study is completely voluntary. You may drop out of this study at any time. Your choice to drop out of this study will not in any way affect your medical treatment from your doctor.

Please ask questions about any and every part of this study you do not understand before you sign and date this Informed Consent Form. If you drop out of the study you cannot re-enter, but this will not affect you in any other way.

If you decide to leave this study after you receive a study shot or are asked to leave by your study doctor, you will be asked to stay in the study to take part in only the safety tests for all remaining study visits and phone calls, or, if you refuse that, to come back to the study doctor's office one last time for safety tests (see Section 4 of this Informed Consent Form). These safety tests and follow up phone calls are to identify any unexpected side effects. Your study doctor will make sure your regular medicines are working if you were on previous medicines. Your study doctor will record your medical condition at the time you leave the study.

#### 11 NEW INFORMATION

You will be told in a timely manner by your study doctor of any new important information about this study, AV7909 study vaccine and BioThrax vaccine, and other therapies that may affect your health, welfare, or willingness to stay in the study. You may be asked to sign and date a new (revised) Informed Consent Form to show that you have been told of this new information. You may contact the study doctor at any time after your participation ends to find out if any new information about this study has become available.

#### 12 STUDY DISCONTINUATION

Your study doctor, the study sponsor (Emergent), or FDA may decide to take you out of the study, without your consent, if it is in your best interest, if the IRB suspends/terminates study approval, if you are unable to meet the requirements of the study, or if the study is cancelled. You may be asked to leave the study if you do not follow study requirements or if the study shows signs of causing medical harm to you. Also, the study sponsor may decide to end the study at any time for any reason.

#### 13 WHOM TO CONATCT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study, please contact the Investigator at the telephone number listed on the first page of this consent document. If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, and/or concerns or complaints regarding this research study, contact:



Please reference the following number when contacting the Study Subject Adviser:

# STATEMENT OF INFORMED CONSENT

| clinica | I study doctor. A signed and date | d copy must be given to the subject for his/her r | ecords. |
|---|---|---|---|
| Site C | ode: | Subject Identification Number: | |
| Study | Number: | Name of Investigator: | _ |
| You (t | he participant) must complete the | e following: | |
| | | <u>!</u> | Please Tick Boxes |
| 1. | I confirm that I have read this In | formed Consent Form for the above study. | |
| 2. | | n explained to my satisfaction and I have had the questions. I know whom to contact if I think of | |
| 3. | | on is voluntary and that I am free to withdraw at<br>an and without my medical care or legal rights | |
| 4. | individuals appointed by the stu<br>IRB, and regulatory authorities s | medical notes may be looked at by responsible dy sponsor (Emergent), ethics boards, such as the FDA where it is relevant to my taking on for these individuals to have direct access to | ne |
| 5. | | ee to the transfer of my personal data to horities both within and outside the U.S. | |
| 6. | I have been given the information health information from this res | on about the use and disclosure of my protected search. | |
| 7. | By signing and dating this author rights. | rization form, I have not given up any of my legal | |
| 8. | | es of my health information for the purposes isted in this Informed Consent Form for this | |
| 9. | I understand and agree to my pr<br>participation in the study (if app | rimary physician being notified of my<br>dicable). | |
| 10 | . All my questions have been answ | vered. | |
| 11 | . I agree to take part in the above | study. | |

Revised «PIApprovalDate»

«PiFullName»

| | 1 1 | |
|---|---|---|
| Signature of Participant | //////// | hr clock) |
| Print Name of Participant Here | . <u></u> | |
| Retention of blood samples for f | uture use (choose one): | |
| I agree to the storage of my lefto<br>the anthrax vaccine | ver blood samples for future re-testing as | s part of continued research on |
| YES, I agree to allow my blood samples to be retained for future analysis. | Participant's Signature | Date of signature |
| NO, I decline to allow my blood samples to be retained for future analysis. | Participant's Signature | Date of signature |
| Signature of Person Explaining Co | onsent YYYY/MMM/DD Time (24 | hr clock) |
| Print Name of Person Explaining | <br>Consent Here | |
| | the best of my knowledge, the individual tudy fully and carefully explained and clear in this research project. | |
| Signature of Investigator | YYYY/MMM/DD T | ime (24hr clock) |
| Print Name of Investigator Here | | |